CLINICAL TRIAL: NCT00491335
Title: HIV Infection and Tobacco Use Among Injection Drug Users in Baltimore, MD: A Pilot Study of Biomarkers
Brief Title: HIV Infection and Tobacco Use Among Injection Drug Users in Baltimore, Maryland: A Pilot Study of Biomarkers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907173; 07-C-N173
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-02-16

CONDITIONS: HIV Infections; AIDS; Lung Cancer; Tobacco Addiction; Drug Addiction
Keywords: AIDS; Lung Cancer; Emphysema; Nicotine; HIV Infection; Smoking
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Lung Neoplasms; Substance-Related Disorders; Emphysema; Smoking

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

The incidence of lung cancer is quite high among people with the human immunodeficiency (HIV) virus. Frequent smoking may explain that cancer increase, given that 50% to 70% of HIV-infected people are current smokers.

Recent research suggests that other factors may be involved as well. Smoking habits, such as smoking earlier in life or smoking more cigarettes a day than others do, may have a role. Also, HIV-infected smokers seem to have a greater risk of chronic obstructive pulmonary disease (COPD). The association of HIV and COPD is important, because COPD itself is linked to an increased risk of lung cancer.

About 1,600 subjects from the study known as ALIVE (AIDS Linked to the Intra-Venous Experience), which began in 1988 in Baltimore, Maryland, will be given a detailed questionnaire on smoking behaviors and lung cancer risk factors. They will also have spirometry testing, to evaluate lung function.

Objectives:

To better characterize smoking habits and compare tobacco use among HIV-infected and uninfected drug users.

To compare serum cotinine levels and spirometry results, as a marker of tobacco use and a marker of damage to lung function, respectively.

Eligibility:

Patients 18 years of age and older who are in the ALIVE cohort.

Design:

Patients undergo the following procedures:

* Completing a questionnaire on smoking history. Questions include age when smoking began, periods of quitting smoking, average number of cigarettes per day for specific periods, amount of each cigarette smoked, depth of inhalation, type of cigarette, nicotine dependence, use of other smoked [Note: I would not mention that these drugs are illegal] drugs, exposure to environmental tobacco smoke, past medical history, and recent respiratory symptoms.
* Spirometry testing. Patients are asked to breathe as deeply as possible and then rapidly exhale into a tube. The forced expiration volume in 1 second reflects the average flow rate during the first second, and it can be used to determine the degree of pulmonary obstruction.
* Blood samples. Tests measure levels of cotinine, a chemical made by the body from nicotine. African American males, who constitute the majority of the ALIVE cohort, participate in this test. Results would show how much tobacco smoke has recently entered the body. For this test, researchers plan to evaluate 240 current tobacco smokers and 100 participants who report no recent cigarette use.

DETAILED DESCRIPTION:
Lung cancer incidence is substantially elevated among people infected with human immunodeficiency virus (HIV). Although frequent smoking may partly explain this increase, recent work suggests other factors may also be involved. To better characterize smoking habits and lung cancer risk in HIV-infected people, the investigators propose a cross-sectional pilot study of HIV-infected and uninfected injection drug users in the ALIVE cohort in Baltimore, Maryland. A detailed questionnaire on smoking behaviors and other lung cancer risk factors will be administered to all ~ 1600 cohort subjects. In addition, the investigators will measure serum cotinine (a marker of recent smoking intensity) for a sample of 340 African American males from the cohort, stratified on the amount of cigarette use, HIV status, and CD4 count. Spirometry will be performed on the entire group of 1600 subjects, to assess for chronic obstructive pulmonary disease. Differences between HIV-infected and uninfected subjects in smoking habits, exposure to tobacco, or lung damage will identify areas for future investigation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Must be a participant in the ALIVE Study

EXCLUSION CRITERIA:

Not a participant in the ALIVE Study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-06-18; Study Completion 2010-02-16

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Parker MS, Leveno DM, Campbell TJ, Worrell JA, Carozza SE. AIDS-related bronchogenic carcinoma: fact or fiction? Chest. 1998 Jan;113(1):154-61. doi: 10.1378/chest.113.1.154. PMID 9440583
- [Background] Phelps RM, Smith DK, Heilig CM, Gardner LI, Carpenter CC, Klein RS, Jamieson DJ, Vlahov D, Schuman P, Holmberg SD; HER Study Group. Cancer incidence in women with or at risk for HIV. Int J Cancer. 2001 Dec 1;94(5):753-7. doi: 10.1002/ijc.1528. PMID 11745473
- [Background] Hessol NA, Seaberg EC, Preston-Martin S, Massad LS, Sacks HS, Silver S, Melnick S, Abulafia O, Levine AM; WIHS Collaborative Study Group. Cancer risk among participants in the women's interagency HIV study. J Acquir Immune Defic Syndr. 2004 Aug 1;36(4):978-85. doi: 10.1097/00126334-200408010-00013. PMID 15220706